CLINICAL TRIAL: NCT05008224
Title: Phase 2 Study of Pembrolizumab and Chemotherapy in Patients With Newly Diagnosed Classical Hodgkin Lymphoma (KEYNOTE-C11)
Brief Title: Study of Safety and Efficacy of Pembrolizumab and Chemotherapy in Participants With Newly Diagnosed Classical Hodgkin Lymphoma (cHL) (MK-3475-C11/KEYNOTE-C11)
Acronym: KEYNOTE-C11
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 3475-C11; MK-3475-C11 (Other: MSD); KEYNOTE-C11 (Other: MSD); 2022-501615-14-00 (Registry Identifier: EU CT); U1111-1281-5347 (Registry Identifier: UTN); 2021-001244-95 (EudraCT Number)
Record Dates: First submitted 2021-08-13; First posted 2021-08-17 (Actual); Results first posted 2024-10-16 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2025-05

CONDITIONS: Classical Hodgkin Lymphoma
Keywords: Programmed Cell Death 1 (PD-1, PD1); Programmed Cell Death-Ligand 1 (PD-L1, PDL1); Programmed Cell Death-Ligand 2 (PD-L2, PDL2)
MeSH Terms: conditions — Parkinson Disease 4, Autosomal Dominant Lewy Body | interventions — pembrolizumab; Doxorubicin; liposomal doxorubicin; Vinblastine; Dacarbazine; Bleomycin; Etoposide; etoposide phosphate; Cyclophosphamide; Vincristine; Procarbazine; Prednisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Pembrolizumab Monotherapy + AVD Chemotherapy/escBEACOPP Chemotherapy + Pembrolizumab Consolidation (Experimental): After completing Positron Emission Tomography (PET) scan 1 during eligibility screening, participants received pembrolizumab monotherapy intravenous (IV) for three 3-week cycles followed by PET scan 2.
  Participants next received 2 phases of chemotherapy. In chemotherapy phase 1, all participants received doxorubicin in combination with vinblastine & dacarbazine (AVD) IV for two 4-week cycles followed by PET scan 3. In chemotherapy phase 2, participants who were PET scan 3 negative, or positive and age ≥60 years, received up to 4 additional cycles of AVD IV, while participants who were PET scan 3 positive and age <60 years received up to four 3-week cycles of escalated bleomycin in combination with etoposide, doxorubicin, cyclophosphamide, vincristine, procarbazine, & prednisone (escBEACOPP) IV.
  All participants then received pembrolizumab consolidation IV for four 6-week cycles followed by a final PET scan.
  Interventions: Biological: Pembrolizumab; Drug: Doxorubicin; Drug: Vinblastine; Drug: Dacarbazine; Drug: Bleomycin; Drug: Etoposide; Drug: Cyclophosphamide; Drug: Vincristine; Drug: Procarbazine; Drug: Prednisone

INTERVENTIONS:
Biological: Pembrolizumab — 200 mg IV administered on Day 1 of each 3-week cycle for 3 cycles during pembrolizumab monotherapy.
  400 mg IV administered on Day 1 of each 6-week cycle for 4 cycles as pembrolizumab consolidation.
  Other Names: MK-3475; SCH 900475; KEYTRUDA®
Drug: Doxorubicin — 25 mg/m^2 IV administered as part of AVD chemotherapy on Days 1 and 15 of each 4-week cycle for 2 cycles in all participants after PET scan 2 and up to 4 additional cycles after PET scan 3 (participants who are PET scan 3 negative, or positive and ≥60 years of age).
  35 mg/m^2 IV administered as part of escBEACOPP chemotherapy on Day 1 of each 3-week cycle for up to 4 cycles after PET scan 3 (participants who are PET scan 3 positive, <60 years of age).
  Other Names: Adriamycin; DOXIL®; Rubex®
Drug: Vinblastine — 6 mg/m^2 IV administered as part of AVD chemotherapy on Days 1 and 15 of each 4-week cycle for 2 cycles after PET scan 2 (all participants) and up to 4 additional cycles after PET scan 3 (participants who are PET scan 3 negative, or positive and ≥60 years of age).
  Other Names: Alkaban-AQ®; Velban®
Drug: Dacarbazine — 375 mg/m^2 IV administered as part of AVD chemotherapy on Days 1 and 15 of each 4-week cycle for 2 cycles after PET scan 2 (all participants) and up to 4 additional cycles after PET scan 3 (participants who are PET scan 3 negative, or positive and ≥60 years of age).
  Other Names: Dtic-Dome®
Drug: Bleomycin — 10 units/m^2 IV administered as part of escBEACOPP chemotherapy on Day 8 of each 3-week cycle for up to 4 cycles after PET scan 3 (participants who are PET scan 3 positive and <60 years of age).
  Other Names: Blenoxane®
Drug: Etoposide — 200 mg/m^2 IV administered as part of escBEACOPP chemotherapy on Days 1-3 of each 3-week cycle for up to 4 cycles after PET scan 3 (participants who are PET scan 3 positive and <60 years of age).
  Other Names: Toposar®; VePesid®; Etopophos®; VP-16; Etoposide phosphate
Drug: Cyclophosphamide — 1250 mg/m^2 IV administered as part of escBEACOPP chemotherapy on Day 1 of each 3-week cycle for up to 4 cycles after PET scan 3 (participants who are PET scan 3 positive and <60 years of age).
  Other Names: Neosar®; Cytoxan®
Drug: Vincristine — 1.4 mg/m^2 IV administered as part of escBEACOPP chemotherapy on Day 8 of each 3-week cycle for up to 4 cycles after PET scan 3 (participants who are PET scan 3 positive and <60 years of age).
  Other Names: Oncovin®; Vincasar PFS®
Drug: Procarbazine — 100 mg/m^2 orally (PO) administered as part of escBEACOPP chemotherapy on Days 1-7 of each 3-week cycle for up to 4 cycles after PET scan 3 (participants who are PET scan 3 positive and <60 years of age).
  Other Names: Matulane®
Drug: Prednisone — 40 mg/m^2 PO administered as part of escBEACOPP chemotherapy on Days 1-14 of each 3-week cycle for up to 4 cycles after PET scan 3 (participants who are PET scan 3 positive and <60 years of age).
  Other Names: Liquid Pred®; Meticorten®; Orasone®; Deltasone®

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of pembrolizumab (MK-3475) monotherapy, followed by chemotherapy, followed by pembrolizumab consolidation. The primary hypothesis of the study is that the complete response (CR) rate at the end of study intervention according to Lugano 2014 response criteria is higher than conventional chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

The main inclusion criteria include, but are not limited to the following:

* Has a histologically confirmed diagnosis of Ann Arbor Stage III or IV classical Hodgkin Lymphoma (cHL). Stage I and II participants may be enrolled, but must have at least one National Comprehensive Cancer Network (NCCN) unfavorable risk factor per protocol
* Has measurable 2-fluorodeoxyglucose (FDG)-avid disease based on investigator assessment according to Lugano 2014 response criteria
* Has not received prior radiation therapy, chemotherapy, immunotherapy, or other systemic therapy for the treatment of cHL before the first dose of study intervention
* Has an Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 to 1 assessed within 7 days before the start of study intervention

Exclusion Criteria:

The main exclusion criteria include, but are not limited to the following:

* Has confirmed nodular lymphocyte-predominant Hodgkin Lymphoma (HL)
* Has an uncontrolled intercurrent cardiovascular illness
* Has received prior therapy with an anti-programmed cell death 1 protein (PD-1), anti-programmed cell death ligand 1 protein (PD-L1), or anti- programmed cell death ligand 2 protein (PD-L2) agent or with an agent directed to another stimulatory or coinhibitory T-cell receptor
* Has received or is expected to receive a live or live-attenuated vaccine within 30 days before the first dose of study intervention
* Is currently participating in or has participated in a study of an investigational agent or has used an investigational device within 4 weeks before the first dose of study intervention
* Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior the first dose of study medication
* Has a known additional malignancy that is progressing or has required active treatment within the past 5 years
* Has radiographically detectable central nervous system metastases and/or carcinomatous meningitis
* Has an active autoimmune disease that has required systemic treatment in past 2 years
* Has a history of (noninfectious) pneumonitis/interstitial lung disease that required steroids or has current pneumonitis/interstitial lung disease
* Has a history or current evidence of pulmonary fibrosis
* Has had an allogenic tissue/solid organ transplant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 146 (Actual)
Dates: Start 2021-10-07 (Actual); Primary Completion 2023-10-11 (Actual); Study Completion 2024-05-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (48):
- United States (6):
  - St Joseph Heritage Healthcare-Oncology ( Site 0004), Fullerton, California
  - Stanford Cancer Center ( Site 0023), Palo Alto, California
  - Northwestern Memorial Hospital ( Site 0002), Chicago, Illinois
  - OptumCare Cancer Care-Research Department ( Site 0005), Las Vegas, Nevada
  - University of Tennessee Medical Center-Cancer Institute ( Site 0006), Knoxville, Tennessee
  - Texas Oncology-Plano East ( Site 0020), Plano, Texas
- Australia (5):
  - Liverpool Hospital-Haematology ( Site 0906), Liverpool, New South Wales
  - Mater Misericordiae Limited ( Site 0904), Brisbane, Queensland
  - Princess Alexandra Hospital-Division of Cancer Services Trials Unit ( Site 0907), Woolloongabba, Queensland
  - Monash Health-Haematology Research ( Site 0908), Clayton, Victoria
  - Peter MacCallum Cancer Centre ( Site 0905), Melbourne, Victoria
- Canada (5):
  - Cross Cancer Institute ( Site 0207), Edmonton, Alberta
  - Centre Intégré de Santé et de Services Sociaux de la Montérégie-Centre ( Site 0205), Greenfield Park, Quebec
  - Jewish General Hospital ( Site 0200), Montreal, Quebec
  - McGill University Health Centre ( Site 0209), Montreal, Quebec
  - Hopital du Sacre-Coeur de Montreal ( Site 0206), Montreal, Quebec
- Chile (5):
  - Instituto Nacional del Cancer ( Site 1205), Chile, Region M. de Santiago
  - FALP-UIDO ( Site 1202), Santiago, Region M. de Santiago
  - Clínica Alemana de Santiago ( Site 1206), Santiago, Region M. de Santiago
  - Pontificia Universidad Catolica de Chile-Hemato-Oncology ( Site 1204), Santiago, Region M. de Santiago
  - Centro Investigación del Cáncer James Lind ( Site 1200), Temuco, Región de la Araucanía
- France (5):
  - CHU Bordeaux Haut-Leveque ( Site 1505), Pessac, Aquitaine
  - Centre Hospitalier Universitaire de Rennes - Hôpital Pontchaillou-haematology ( Site 1502), Rennes, Brittany Region
  - Centre Hospitalier Universitaire Dijon Bourgogne - Hôpital François Mitterrand ( Site 1504), Dijon, Cote-d Or
  - centre hospitalier lyon sud-Service Hématologie ( Site 1501), Pierre-Bénite, Rhone
  - Centre de Lutte Contre le Cancer - Centre Henri Becquerel Normandie Rouen-Service d'Hématologie ( Si, Rouen, Seine-Maritime
- Israel (6):
  - Rambam Health Care Campus ( Site 1907), Haifa
  - Bnai Zion Medical Center-Hematology ( Site 1909), Haifa
  - Hadassah Medical Center ( Site 1901), Jerusalem
  - Sheba Medical Center-Hemato Oncology ( Site 1904), Ramat Gan
  - ZIV Medical Center ( Site 1908), Safed
  - Sourasky Medical Center ( Site 1905), Tel Aviv
- Italy (4):
  - Azienda Ospedaliera Spedali Civili di Brescia-Hemathology ( Site 1801), Brescia, Lombardy
  - ASST Grande Ospedale Metropolitano Niguarda ( Site 1803), Milan, Milano
  - Policlinico S. Orsola- Malpighi-Istituto di Ematologia L. e A. Seragnoli ( Site 1800), Bologna
  - Fondazione Policlinico Universitario Agostino Gemelli-ISTITUTO DI EMATOLOGIA ( Site 1804), Roma
- Poland (4):
  - Klinika Hematologii - Instytut Hematologii i Transfuzjologii-Klinika Hematologii ( Site 0402), Warsaw, Masovian Voivodeship
  - Narodowy Instytut Onkologii im. Marii Sklodowskiej-Curie - Panstwowy Instytut Badawczy w Warszawie (, Warsaw, Masovian Voivodeship
  - Szpital Wojewódzki w Opolu-Hematology Department ( Site 0401), Opole, Opole Voivodeship
  - Uniwersyteckie Centrum Kliniczne-Klinika Hematologii i Transplantologii ( Site 0403), Gdansk, Pomeranian Voivodeship
- Russia (3):
  - Moscow City Clinical Hospital S.P. Botkin ( Site 0702), Moscow, Moscow
  - First Pavlov State Medical University of Saint Petersburg-Raisa Gorbacheva Memorial Institut for Pe, Saint Petersburg, Sankt-Peterburg
  - Almazov National Medical Research Centre ( Site 0704), Saint Petersburg, Sankt-Peterburg
- Spain (2):
  - Instituto Catalan de Oncologia - Hospital Duran i Reynals-Haematology Department ( Site 1031), L'Hospitalet Del Llobregat, Barcelona
  - Hospital Universitario 12 de Octubre ( Site 1032), Madrid
- Turkey (Türkiye) (3):
  - Dokuz Eylül Üniversitesi ( Site 5002), Balçova, İzmir
  - Ankara University Hospital Cebeci-hematology ( Site 5000), Ankara
  - Vehbi Koc Vakfi - Amerikan Hastanesi ( Site 5001), Istanbul

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com/
- See also: Plain Language Summary — https://msd.trialsummaries.com/Study/StudyDetails?id=26282&tenant=MT_MSD_9011

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Male or female participants with newly diagnosed early unfavorable or advanced-stage classical Hodgkin Lymphoma (cHL), who were at least 18 years old, were enrolled in this study.
Pre-assignment Details: 146 participants were allocated to the treatment arm and received sequential treatments beginning with pembrolizumab monotherapy, followed by chemotherapy (phases 1 and 2), and finishing with pembrolizumab consolidation.
  Per protocol, efficacy analysis was planned and conducted on the treatment arm of participants that received these sequential treatments. Safety outcome measures were analyzed based on the individual study treatment received by the participant at the time of the event.
Period: Overall Study
Arm/Group | Pembrolizumab Monotherapy + AVD Chemotherapy/escBEACOPP Chemotherapy + Pembrolizumab Consolidation
Started | 146
Received ≥1 Dose of Pembrolizumab | 146
Received at ≥1 Dose of AVD Chemotherapy | 136
Received at ≥1 Dose of escBEACOPP Chemotherapy | 17
Completed | 0
Not Completed | 146
Not completed — Death | 3
Not completed — Lost to Follow-up | 2
Not completed — Did Not Continue on Extension Study | 39
Not completed — Transferred to Extension Study | 100
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Population: The analysis population consisted of all participants who received at least 1 dose of pembrolizumab
Groups:
- Pembrolizumab Monotherapy + AVD Chemotherapy/escBEACOPP Chemotherapy + Pembrolizumab Consolidation: After completing PET scan 1 during eligibility screening, participants received pembrolizumab monotherapy IV for three 3-week cycles followed by PET scan 2.
  Participants next received 2 phases of chemotherapy. In chemotherapy phase 1, all participants received AVD IV for two 4-week cycles followed by PET scan 3. In chemotherapy phase 2, participants who were PET scan 3 negative, or positive and age ≥60 years, received up to 4 additional cycles of AVD IV, while participants who were PET scan 3 positive and age <60 years received up to four 3-week cycles of escBEACOPP IV.
  All participants then received pembrolizumab consolidation IV for four 6-week cycles followed by a final PET scan.
Arm/Group | Pembrolizumab Monotherapy + AVD Chemotherapy/escBEACOPP Chemotherapy + Pembrolizumab Consolidation
Number analyzed (Participants) | 146
Age, Continuous [Mean (Standard Deviation); unit: Years] | 38.9 (16.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 66
  Male | 80
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 22
  Not Hispanic or Latino | 108
  Unknown or Not Reported | 16
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3
  Asian | 8
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 126
  More than one race | 1
  Unknown or Not Reported | 8

OUTCOME MEASURES:

1. Primary Outcome: Complete Response (CR) Rate at the End of Study Intervention as Assessed by Blinded Independent Central Review (BICR) Per Lugano 2014 Response Criteria
Description: CR rate was assessed by BICR using Computed Tomography (CT) and PET scan according to Lugano 2014 response criteria (Cheson, B.D. et al, Journal of Clinical Oncology, 2014). At each timepoint, CR was determined by combining the anatomic response, metabolic response, and clinical data. The criteria for CR included complete metabolic (no/minimal 2-fluorodeoxyglucose [FDG] uptake) and radiologic response (target lesions regress to ≤1.5 cm in longest transverse diameter of a lesion) and no new lesions. Per protocol, participants who discontinued study intervention during pembrolizumab monotherapy, chemotherapy, or pembrolizumab consolidation, or are lost to follow-up, or receive any new non-study anticancer therapy prior to end of treatment were classified as non-responders. The percentage of participants who had CR after the completion of pembrolizumab consolidation is presented.
Time Frame: Up to approximately 24 months
Population: The analysis population consisted of all participants who received at least 1 dose of pembrolizumab.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Groups:
- Pembrolizumab Monotherapy + AVD Chemotherapy/escBEACOPP Chemotherapy + Pembrolizumab Consolidation: Participants received pembrolizumab monotherapy IV for three 3-week cycles followed by PET scan 2.
  Participants next received 2 phases of chemotherapy. In chemotherapy phase 1, all participants received AVD IV for two 4-week cycles followed by PET scan 3. In chemotherapy phase 2, participants who were PET scan 3 negative, or positive and age ≥60 years, received up to 4 additional cycles of AVD IV, while participants who were PET scan 3 positive and age <60 years received up to four 3-week cycles of escBEACOPP IV.
  All participants then received pembrolizumab consolidation IV for four 6-week cycles followed by a final PET scan.
Arm/Group | Pembrolizumab Monotherapy + AVD Chemotherapy/escBEACOPP Chemotherapy + Pembrolizumab Consolidation
Number analyzed (Participants) | 146
Percentage of Participants | 67.0 [58.9 to 74.7]

2. Secondary Outcome: CR Rate at the End of Study Intervention as Assessed by Investigator Per Lugano 2014 Response Criteria
Description: CR rate was assessed by the investigator using CT and PET scan according to Lugano 2014 response criteria (Cheson, B.D. et al, Journal of Clinical Oncology, 2014). At each timepoint, CR was determined by combining the anatomic response, metabolic response, and clinical data. The criteria for CR included complete metabolic (no/minimal FDG uptake) and radiologic response (target lesions regress to ≤1.5 cm in longest transverse diameter of a lesion) and no new lesions. Per protocol, participants who discontinued study intervention during pembrolizumab monotherapy, chemotherapy, or pembrolizumab consolidation, or are lost to follow-up, or receive any new non-study anticancer therapy prior to end of treatment were classified as non-responders. The percentage of participants who had CR after the completion of pembrolizumab consolidation is presented.
Time Frame: Up to approximately 31 months
Population: The analysis population consisted of all participants who received at least 1 dose of pembrolizumab.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Pembrolizumab Monotherapy + AVD Chemotherapy/escBEACOPP Chemotherapy + Pembrolizumab Consolidation
Number analyzed (Participants) | 146
Percentage of Participants | 71.9 [63.9 to 79.0]

3. Secondary Outcome: Duration of Complete Response (DurCR) as Assessed by BICR Per Lugano 2014 Response Criteria
Description: DurCR was defined as the time from CR to progressive disease (PD) or death due to any cause, whichever came first. CR was assessed by BICR using CT and PET scan according to Lugano 2014 response criteria (Cheson, B.D. et al, Journal of Clinical Oncology, 2014). At each timepoint, CR was determined by combining the anatomic response, metabolic response, and clinical data. The criteria for CR included complete metabolic (no/minimal FDG uptake) and radiologic response (target lesions regress to ≤1.5 cm in longest transverse diameter of a lesion) and no new lesions. PD was defined as uptake moderately or markedly higher than the liver and/or new lesions. DurCR was analyzed by the Kaplan-Meier method for censored data and is presented for participants who demonstrated CR.
Time Frame: Up to approximately 31 months
Population: The analysis population consisted of all participants who received at least 1 dose of pembrolizumab and who had achieved CR.
  DurCR data was censored on the date of the last disease assessment documenting absence of PD for participants who do not have progression and are still on study at the time of an analysis, are given antitumor treatment other than the study treatment, or are removed from study prior to documentation of tumor progression.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab Monotherapy + AVD Chemotherapy/escBEACOPP Chemotherapy + Pembrolizumab Consolidation
Number analyzed (Participants) | 121
Months | NA [NA to NA] — NA = Median DurCR and upper and lower 95% confidence limits not reached at time of data cut-off due to an insufficient number of responding participants with relapse.

4. Secondary Outcome: Rate of PET Negativity Assessed by BICR According to the FDG-PET 5-point Scale After Administration of Pembrolizumab Monotherapy (PET Scan 2)
Description: The rate of PET negativity was defined as the percentage of participants considered negative on the FDG-PET 5-point scale, as assessed by BICR according to Lugano 2014 response criteria (Cheson, B.D. et al, Journal of Clinical Oncology, 2014). Participants were assigned a single score on the FDG-PET 5-point scale measuring FDG uptake (1 = no uptake above background, 2 = uptake above background but ≤ mediastinum, 3 = uptake > mediastinum but ≤ liver, 4 = uptake moderately > liver, 5 = uptake markedly > liver or new FDG-positive lesions). Higher scores corresponded to greater uptake (greater disease). FDG-PET 5-point scale scores of 1, 2, and 3 were considered negative and scores of 4 and 5 were considered positive. The percentage of participants who were assessed as negative at PET scan 2, after completion of 3 cycles of pembrolizumab monotherapy, is presented.
Time Frame: Up to approximately 10 weeks
Population: The analysis population consisted of all participants who had completed 3 cycles of pembrolizumab monotherapy.
Measure: Number; unit: Percentage of Participants
Groups:
- Pembrolizumab Monotherapy: Participants received pembrolizumab monotherapy IV for three 3-week cycles followed by PET scan 2.
Arm/Group | Pembrolizumab Monotherapy
Number analyzed (Participants) | 146
Percentage of Participants | 19.9

5. Secondary Outcome: Rate of PET Negativity Assessed by BICR According to the FDG-PET 5-point Scale After Administration of Pembrolizumab Monotherapy and AVD Chemotherapy (PET Scan 3)
Description: The rate of PET negativity was defined as the percentage of participants considered negative on the FDG-PET 5-point scale, as assessed by BICR according to Lugano 2014 response criteria (Cheson, B.D. et al, Journal of Clinical Oncology, 2014). Participants were assigned a single score on the FDG-PET 5-point scale measuring FDG uptake (1 = no uptake above background, 2 = uptake above background but ≤ mediastinum, 3 = uptake > mediastinum but ≤ liver, 4 = uptake moderately > liver, 5 = uptake markedly > liver or new FDG-positive lesions). Higher scores corresponded to greater uptake (greater disease). FDG-PET 5-point scale scores of 1, 2, and 3 were considered negative and scores of 4 and 5 were considered positive. The percentage of participants who were assessed as negative at PET scan 3, after completion of 3 cycles of pembrolizumab monotherapy and phase 1 AVD chemotherapy (2 AVD cycles), is presented.
Time Frame: Up to approximately 5 months
Population: The analysis population consisted of all participants who had completed 3 cycles of pembrolizumab monotherapy and phase 1 AVD chemotherapy (2 AVD cycles).
Measure: Number; unit: Percentage of Participants
Groups:
- Pembrolizumab Monotherapy + AVD Chemotherapy: Participants received pembrolizumab monotherapy IV for three 3-week cycles.
  Next, in chemotherapy phase 1, all participants received AVD IV for two 4-week cycles followed by PET scan 3.
Arm/Group | Pembrolizumab Monotherapy + AVD Chemotherapy
Number analyzed (Participants) | 146
Percentage of Participants | 70.5

6. Secondary Outcome: Number of Participants Who Experienced an Adverse Event (AE)
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a study intervention. Per protocol, collection and reporting of AEs was based on the study treatment received by the participant (pembrolizumab, AVD chemotherapy, or escBEACOPP chemotherapy) at the time of the event. The number of participants who experienced an AE is reported.
Time Frame: Up to approximately 31 months
Population: The analysis population consisted of all participants who received at least 1 dose of study intervention. Per protocol, analysis was based on the study treatment received by the participant (pembrolizumab, AVD chemotherapy, or escBEACOPP chemotherapy) at the time of the event.
Measure: Count of Participants; unit: Participants
Groups:
- Pembrolizumab Monotherapy and Consolidation: Participants received pembrolizumab monotherapy IV for three 3-week cycles followed by PET scan 2.
  Participants also receive pembrolizumab consolidation IV for four 6-week cycles followed by a final PET scan.
  Per protocol, collection and reporting of AEs was based on the individual study treatment received by the participant (i.e., pembrolizumab) at the time of the event.
- AVD Chemotherapy: In chemotherapy phase 1, participants received AVD IV for two 4-week cycles followed by PET scan 3. In chemotherapy phase 2, participants who were PET scan 3 negative, or positive and age ≥60 years, received up to 4 additional cycles of AVD IV.
  Per protocol, collection and reporting of AEs was based on the individual study treatment received by the participant (i.e., AVD chemotherapy) at the time of the event.
- escBEACOPP Chemotherapy: In chemotherapy phase 2, participants who were PET scan 3 positive and age <60 years received up to four 3-week cycles of escBEACOPP IV.
  Per protocol, collection and reporting of AEs was based on the individual study treatment received by the participant (i.e., escBEACOPP chemotherapy) at the time of the event.
Arm/Group | Pembrolizumab Monotherapy and Consolidation | AVD Chemotherapy | escBEACOPP Chemotherapy
Number analyzed (Participants) | 146 | 136 | 17
Participants | 135 | 132 | 17

7. Secondary Outcome: Number of Participants Who Discontinued Study Treatment Due to an AE
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a study intervention. Per protocol, collection and reporting of AEs was based on the study treatment received by the participant (pembrolizumab, AVD chemotherapy, or escBEACOPP chemotherapy) at the time of the event. The number of participants who discontinued study intervention due to an AE is reported.
Time Frame: Up to approximately 17 months
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | Pembrolizumab Monotherapy and Consolidation | AVD Chemotherapy | escBEACOPP Chemotherapy
Number analyzed (Participants) | 146 | 136 | 17
Participants | 15 | 1 | 0

ADVERSE EVENTS:
Time Frame: Up to approximately 31 months
Description: All-Cause Mortality included all allocated participants. Serious and Other AEs included all participants who received ≥1 dose of study intervention. As pre-specified by the protocol, MedDRA preferred terms "Neoplasm progression", "Malignant neoplasm progression" and "Disease progression" that were not related to study drug were excluded as AEs. Per protocol, reporting of All-Cause Mortality and AEs was based on the individual study treatment received by the participant at the time of the event.
Groups:
- Pembrolizumab Monotherapy and Consolidation: Participants received pembrolizumab monotherapy IV for three 3-week cycles followed by PET scan 2. Participants also received pembrolizumab consolidation IV for four 6-week cycles followed by a final PET scan.
  Per protocol, collection and reporting of AEs was based on the individual study treatment received by the participant (i.e., pembrolizumab) at the time of the event.
Arm/Group | Pembrolizumab Monotherapy and Consolidation | AVD Chemotherapy | escBEACOPP Chemotherapy
All-Cause Mortality (participants affected / at risk) | 0/146 | 3/136 | 0/17
Serious Adverse Events (participants affected / at risk) | 26/146 | 26/136 | 6/17
Other Adverse Events (participants affected / at risk) | 122/146 | 131/136 | 17/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pembrolizumab Monotherapy and Consolidation (N=146) | AVD Chemotherapy (N=136) | escBEACOPP Chemotherapy (N=17)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 12 (15) | 3 (7)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (2) | 0 (0) | 0 (0)
Cardiac tamponade (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Chills (General disorders) | 0 (0) | 1 (1) | 0 (0)
Mucosal inflammation (General disorders) | 1 (1) | 2 (4) | 0 (0)
Pyrexia (General disorders) | 6 (6) | 3 (4) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Immune-mediated hepatitis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Cytokine release syndrome (Immune system disorders) | 2 (2) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
COVID-19 (Infections and infestations) | 1 (1) | 2 (2) | 0 (0)
Campylobacter gastroenteritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Device related sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Meningitis aseptic (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Meningitis viral (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Pseudomonas infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Rhinovirus infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Sialoadenitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Urosepsis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Toxicity to various agents (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Chest wall necrosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Immune-mediated encephalitis (Nervous system disorders) | 3 (3) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pembrolizumab Monotherapy and Consolidation (N=146) | AVD Chemotherapy (N=136) | escBEACOPP Chemotherapy (N=17)
Anaemia (Blood and lymphatic system disorders) | 9 (13) | 19 (26) | 8 (9)
Eosinophilia (Blood and lymphatic system disorders) | 12 (16) | 3 (3) | 1 (1)
Leukopenia (Blood and lymphatic system disorders) | 1 (1) | 8 (17) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 3 (5) | 19 (32) | 3 (3)
Pancytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 4 (4) | 6 (8)
Angina pectoris (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Myocardial ischaemia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 2 (2) | 2 (4) | 2 (2)
Hyperthyroidism (Endocrine disorders) | 15 (16) | 5 (5) | 0 (0)
Hypothyroidism (Endocrine disorders) | 11 (15) | 11 (11) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 7 (7) | 4 (5) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 2 (2) | 10 (14) | 0 (0)
Constipation (Gastrointestinal disorders) | 5 (5) | 34 (47) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 15 (15) | 12 (18) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 3 (3) | 2 (2) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 5 (6) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 (2) | 5 (5) | 2 (2)
Nausea (Gastrointestinal disorders) | 15 (15) | 54 (89) | 3 (3)
Odynophagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Oral pain (Gastrointestinal disorders) | 1 (1) | 6 (16) | 1 (1)
Rectal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (2)
Salivary hypersecretion (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 1 (2) | 6 (7) | 3 (4)
Vomiting (Gastrointestinal disorders) | 3 (3) | 13 (16) | 3 (4)
Asthenia (General disorders) | 5 (5) | 11 (12) | 0 (0)
Chills (General disorders) | 6 (7) | 1 (1) | 1 (1)
Fatigue (General disorders) | 16 (16) | 20 (21) | 4 (4)
Malaise (General disorders) | 0 (0) | 0 (0) | 1 (1)
Mucosal inflammation (General disorders) | 2 (2) | 7 (7) | 6 (7)
Pain (General disorders) | 3 (3) | 2 (2) | 1 (1)
Pyrexia (General disorders) | 31 (35) | 17 (19) | 3 (3)
COVID-19 (Infections and infestations) | 18 (20) | 26 (26) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 11 (12) | 5 (5) | 1 (1)
Accidental overdose (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (2)
Alanine aminotransferase increased (Investigations) | 25 (29) | 15 (17) | 3 (5)
Aspartate aminotransferase increased (Investigations) | 10 (10) | 7 (8) | 2 (3)
Blood alkaline phosphatase increased (Investigations) | 4 (4) | 3 (5) | 2 (2)
Blood bicarbonate decreased (Investigations) | 1 (1) | 1 (1) | 1 (1)
Blood creatinine increased (Investigations) | 2 (2) | 2 (2) | 1 (1)
Blood thyroid stimulating hormone increased (Investigations) | 6 (8) | 2 (3) | 1 (1)
Lymphocyte count decreased (Investigations) | 4 (6) | 11 (19) | 4 (6)
Neutrophil count decreased (Investigations) | 11 (15) | 85 (165) | 7 (12)
Platelet count decreased (Investigations) | 1 (1) | 2 (3) | 3 (5)
Transaminases increased (Investigations) | 2 (2) | 1 (1) | 1 (1)
White blood cell count decreased (Investigations) | 7 (10) | 24 (46) | 6 (11)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1)
Hyperphosphataemia (Metabolism and nutrition disorders) | 2 (2) | 3 (3) | 2 (2)
Hypocalcaemia (Metabolism and nutrition disorders) | 2 (3) | 2 (4) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 3 (3) | 1 (1) | 4 (5)
Hypomagnesaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 1 (1)
Lactic acidosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 13 (18) | 7 (7) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 14 (16) | 3 (3)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (2) | 4 (4) | 2 (2)
Headache (Nervous system disorders) | 19 (20) | 7 (7) | 2 (4)
Neuropathy peripheral (Nervous system disorders) | 4 (4) | 14 (14) | 1 (1)
Paraesthesia (Nervous system disorders) | 1 (1) | 2 (3) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1) | 16 (17) | 1 (2)
Presyncope (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 9 (9) | 7 (7) | 1 (1)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Urinary retention (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 8 (9) | 9 (10) | 2 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 4 (4) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 6 (8) | 10 (11) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 17 (17) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 3 (3) | 1 (1) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 20 (24) | 5 (6) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 11 (13) | 6 (6) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 9 (11) | 1 (1) | 2 (3)
Hypotension (Vascular disorders) | 3 (3) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The results of this study may be published or presented at scientific meetings. The Sponsor will generally support publication of multicenter studies only in their entirety and not as individual site data. If publication activity is not directed by the Sponsor, the investigator agrees to submit all manuscripts or abstracts to the Sponsor before submission. Authorship will be determined by mutual agreement and in line with International Committee of Medical Journal Editors requirements.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-12-15): https://cdn.clinicaltrials.gov/large-docs/24/NCT05008224/Prot_SAP_001.pdf